CLINICAL TRIAL: NCT00244348
Title: Hepatic Arterial Infusion of Oxaliplatin Clinical Trial
Brief Title: Hepatic Artery Infusion With Oxaliplatin
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator has left institution
Sponsor: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRRC#341-05
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Cancer; Metastasis; Liver Cancer
Keywords: hepatic artery infusion; colorectal cancer; liver metastasis; oxaliplatin; 5 fluorouracil
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms | interventions — Oxaliplatin; Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin (via HAI)
Drug: 5 Fluorouracil (systemic)

SUMMARY:
Hepatic artery infusion (HAI) with oxaliplatin (OX), systemic 5 fluorouracil (5FU), and leucovorin (HAI/OX/FU) will be implemented using an interventional radiology technique to obviate the need for initial major surgery (catheter placement) in patients who have unresectable liver metastasis from colorectal cancer. The study goal is to reduce tumor size to make possible a complete resection of all lesions. Secondary goals are to reduce or eliminate the complexity usually associated with HAI, to accomplish most or all of the treatment as an outpatient, to reduce costs, and to avoid the hepatotoxicity associated with HAI/floxuridine (FUDR). Oxaliplatin has been selected because of its ease of use, known toxicology, and established efficacy in colorectal cancer.

DETAILED DESCRIPTION:
After entry qualification and registration patients will undergo hepatic artery catheterization via interventional radiology. The catheter will remain in place for two hours while oxaliplatin is infused and then be removed. This treatment will be followed by a 48 hour infusion of 5FU and leucovorin, generally following the principle of FOLFOX 6. These cycles of therapy will be repeated biweekly for six episodes. Hepatic tumor size will be evaluated by CT scan to determine if resectability has been established as the result of tumor size reduction. If so, the patient will be offered resection of the residual lesions in an effort to achieve long term survival.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent
2. Age greater than 17 years
3. Stage IV colorectal cancer
4. Metastasis limited to the liver considered unresectable for cure by standard methods
5. Completely resected primary tumor
6. Life expectancy greater than 3 years excluding cancer
7. Eastern Cooperative Oncology Group (ECOG) status 0, 1, 2
8. Absolute granulocyte count greater than 1500
9. Platelet count greater than 100,000
10. Adequate hepatic function
11. Adequate renal function

Exclusion Criteria:

1. Concomitant anticancer therapy other than this protocol
2. Gastroduodenal ulcer
3. Pregnancy or lactation
4. Last treatment for colon cancer less than 4 weeks from this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
number of patients who become eligible for total resection of metastatic liver tumor
overall survival of patients resected for cure versus (vs.) resected for palliation vs. not resected.

SECONDARY OUTCOMES:
toxicity
HAI complexity
cost

CONTACTS AND LOCATIONS:
Overall Officials: Robert K Ausman, M. D., Principal Investigator — Dept. Surgery, Medical College of Wisconsin; Edward J Quebbeman, M. D., Principal Investigator — Dept. Surgery, Medical College of Wisconsin; William S Rilling, M. D., Principal Investigator — Dept. Radiology, Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/ Froedtert Hospital, Milwaukee, Wisconsin, United States